CLINICAL TRIAL: NCT04359771
Title: Yellow Micropulse Laser 577-nm vs Infrared Diode Micropulse Laser 810-nm for the Treatment of Diabetic Macular Edema
Brief Title: Transfoveal Micropulse Laser for Center Involving Diabetic Macular Edema
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelbaki, lecturer of ophthalmology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I-030416
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Results first posted 2020-06-01 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Diabetic Retinopathy; Macula Edema
Keywords: micro-pulse laser; trans-foveal
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Yellow MPL (Active Comparator)
  Interventions: Device: Yellow micro-pulse laser
- Diode MPL (Active Comparator)
  Interventions: Device: Diode micro-pulse laser

INTERVENTIONS:
Device: Yellow micro-pulse laser — applying 577-nm yellow laser in a micro-pulse mode over the macular area including the fovea
  Arms: Yellow MPL
Device: Diode micro-pulse laser — applying 810-nm infra-red diode laser in a micro-pulse mode over the macular area including the fovea
  Arms: Diode MPL

SUMMARY:
Anti-vascular endothelial growth factor (VEGF) therapy is currently the mainstay of treatment for diabetic macular edema (DME). One of the main obstacles of anti-VEGF therapy is the need of repeated injections, which carries both economic and compliance problems to the patients.there is a growing evidence that recognises the effectiveness of the use of micropulse laser (MPL) in treatment of DME. with MPL, it is possible to deliver a subthreshold laser that is above the threshold of biochemical effect but below the threshold of a visible, destructive lesion thereby preventing collateral damage.The MPL technique is available at near - infrared 810 nm diode laser (diode MPL) and at 577 nm (yellow MPL). The current study was conducted in order to compare the efficacy of both MPL techniques in the treatment of center involving DME.

DETAILED DESCRIPTION:
This was a prospective randomized comparative study that included 30 eyes of 15 patients with bilateral DME. The patients were recruited from the Retina Clinic at Kasr Al Ainy Hospital, Cairo University. The study's protocol was reviewed and approved by board of the ophthalmology department, Cairo University, and was in concordance with the tents of Declaration of Helsinki. Eligible patients were informed about the study's objectives, methodology, risks and benefits. A written informed consent was obtained from every patient included in this study.Preliminary examination was in the form of slit-lamp examination, fundus examination, intra ocular pressure measurement, and best corrected visual acuity (BCVA) measurement. A spectral domain optical coherence tomogram (OCT) scan was performed to all patients before treatment to measure the central retinal thickness (CRT). The eyes were randomized into two groups; one eye (right eye) of each patient was treated with 577-nm yellow MPL and the other eye (left eye) of the same patient with Infrared 810-nm diode MPL. Changes in the BCVA and CRT were measured after treatment at 1 and 3 months of follow up.

ELIGIBILITY:
Inclusion Criteria:

* bilateral diabetic macular edema
* center involving confirmed by Optical coherence tomogram (OCT)

Exclusion Criteria:

* any non-diabetic macular edema
* significant media opacities
* previous laser treatment, any intraocular surgery within the past 6 months
* previous intravitreal injections of any drug within the past 6 months

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2018-09-25 (Actual); Study Completion 2018-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hany S Hamza, MD, Study Director — Cairo University
Locations (1):
- Faculty of Medicine, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: starting 6 months after publication
Access Criteria: Individual participant data (IPD) can be shared with researchers who are planning to conduct a similar study. Requests can be sent to the central contacts by email

REFERENCES:
- [Background] Vujosevic S, Martini F, Longhin E, Convento E, Cavarzeran F, Midena E. SUBTHRESHOLD MICROPULSE YELLOW LASER VERSUS SUBTHRESHOLD MICROPULSE INFRARED LASER IN CENTER-INVOLVING DIABETIC MACULAR EDEMA: Morphologic and Functional Safety. Retina. 2015 Aug;35(8):1594-603. doi: 10.1097/IAE.0000000000000521. PMID 25719988
- [Background] Scholz P, Altay L, Fauser S. A Review of Subthreshold Micropulse Laser for Treatment of Macular Disorders. Adv Ther. 2017 Jul;34(7):1528-1555. doi: 10.1007/s12325-017-0559-y. Epub 2017 May 24. PMID 28540655

RESULTS

PARTICIPANT FLOW:
Recruitment Details: one eye (Right) from each patient was assigned to one arm (yellow MPL) and the other eye (Left) of the same patient to the 2nd arm (diode MPL). Therefore, the total number of enrolled participants was 15 contributing to total of 30 eyes (units) i.e there were 15 participants contributing to 15 eyes in each arm of the study.
Units Other Than Participants: eyes
Groups:
- Yellow MPL: Yellow micro-pulse laser: applying 577-nm yellow laser in a micro-pulse mode over the macular area including the fovea. One eye (right) of each participant was assigned to this group.
- Diode MPL: Diode micro-pulse laser: applying 810-nm infra-red diode laser in a micro-pulse mode over the macular area including the fovea. One eye (left) of each participant was assigned to this group.
Period: Overall Study
Arm/Group | Yellow MPL | Diode MPL
Started (1 eye from each patient was assigned to one arm and the other eye of the same patient to the 2nd arm) | 15; 15 eyes (Right eye of every participant was assigned to the diode MPL group) | 15; 15 eyes (Left eye of every participant was assigned to the diode MPL group)
Completed (1 eye from each patient was assigned to one arm and the other eye of the same patient to the 2nd arm) | 13; 13 eyes (The right eye of each participant was assigned to the diode MPL group) | 13; 13 eyes (The left eye of every participant was assigned to the diode MPL group)
Not Completed | 2; 2 eyes | 2; 2 eyes
Not completed — Lack of Efficacy | 2 | 2

BASELINE CHARACTERISTICS:
Population: there were 15 enrolled participants, then two were excluded due to lack of efficacy. So, the analysis population was 13 participants contributing 26 units (eyes).
Groups:
- Total: Total of all reporting groups
Arm/Group | Yellow MPL | Diode MPL | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: two participants were excluded due to lack of efficacy.
  years | 58.23 (8.03) | 58.23 (8.03) | 58.23 (8.03)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: two participants were excluded due to lack of efficacy.
  Participants
    Female | 5 | 5 | 10
    Male | 8 | 8 | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — Population: two participants were excluded due to lack of efficacy
  participants
    Egypt | 13 | 13 | 13

OUTCOME MEASURES:

1. Primary Outcome: Change in Central Retinal Thickness (CRT)
Description: detecting changes in the thickness of the center of the macula
Time Frame: baseline, at 1 month and 3 months after the intervention
Measure: Mean (Standard Deviation); unit: micrometer
Units Other Than Participants: eyes
Arm/Group | Yellow MPL | Diode MPL
Number analyzed (Participants) | 13 | 13
Number analyzed (eyes) | 13 | 13
micrometer
  Baseline | 384.62 (147.06) | 374 (130.42)
  1 month | 349.15 (141.78) | 357.62 (116.23)
  3 months | 321.92 (126.65) | 339.69 (111.94)

2. Primary Outcome: Change in the Best Corrected Visual Acuity (BCVA)
Description: detecting changes in the the best corrected visual acuity in logMAR. A LogMAR chart comprises rows of letters and is used by ophthalmologists, optometrists and vision scientists to estimate visual acuity. This chart was developed at the National Vision Research Institute of Australia in 1976, and is designed to enable a more accurate estimate of acuity than do other charts (e.g., the Snellen chart). For this reason, the LogMAR chart is recommended, particularly in a research setting. A Snellen score of 6/6 (20/20), indicating that an observer can resolve details as small as 1 minute of visual angle, corresponds to a LogMAR of 0 (since the base-10 logarithm of 1 is 0); a Snellen score of 6/12 (20/40), indicating an observer can resolve details as small as 2 minutes of visual angle, corresponds to a LogMAR of 0.3 (since the base-10 logarithm of 2 is near-approximately 0.3), and so on.Therefore, a higher logMAR scores mean a worse outcome.
Time Frame: baseline, at 1 month and 3 months after the intervention
Measure: Mean (Standard Deviation); unit: logMar
Units Other Than Participants: eyes
Arm/Group | Yellow MPL | Diode MPL
Number analyzed (Participants) | 13 | 13
Number analyzed (eyes) | 13 | 13
logMar
  Baseline | 0.68 (0.30) | 0.58 (0.28)
  1 month | 0.60 (0.33) | 0.57 (0.29)
  3 months | 0.55 (0.34) | 0.52 (0.31)

ADVERSE EVENTS:
Time Frame: data were collected over 6 months
Description: the interventions used in the trial are localized to the eye with no systemic complications. in addition, no ocular serious events were reported
Arm/Group | Yellow MPL | Diode MPL
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-12-10): https://cdn.clinicaltrials.gov/large-docs/71/NCT04359771/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-10): https://cdn.clinicaltrials.gov/large-docs/71/NCT04359771/SAP_001.pdf